CLINICAL TRIAL: NCT04411537
Title: A Phase II Trial of Immunotherapy Combined With Neoadjuvant Chemoradiotherapy in Microsatellite Stable Locally Advanced Rectal Cancer
Brief Title: The Combination of Immunotherapy and Neoadjuvant Chemoradiotherapy in MSS Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2019-97-1731
Record Dates: First submitted 2020-05-10; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — spartalizumab; Capecitabine; Irinotecan; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A total of 50 MSS LARC patients will receive 2 cycles of PD-1 antibody, followed by capecitabine plus irinotecan radiosensitized neoadjuvant chemoradiotherapy, and another 3 cycles of PD-1 antibody, finally received the total mesorectal excision (TME) and 6 cycles of adjuvant chemotherapy of XELOX.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: Irinotecan; Radiation: Neoadjuvant Radiotherapy

INTERVENTIONS:
Drug: PD-1 antibody — Before neo-CRT: 2 cycles of PD-1 antibody, 240mg d1 q2w. After neo-CRT: 3 cycles of PD-1 antibody, 240mg d1 q2w.
Drug: Capecitabine — During neo-CRT: 625mg/m2 bid Monday-Friday per week
  Other Names: Xeloda
Drug: Irinotecan — During neo-CRT: 80mg/m2 qw (UGT1A1*28 6/6) or 65mg/m2 qw (UGT1A1*28 6/7)
Radiation: Neoadjuvant Radiotherapy — IMRT DT: 50Gy/25Fx

SUMMARY:
The study evaluates the addition of immunotherapy of PD-1 antibody in neoadjuvant chemoradiotherapy in microsatellite stable (MSS) locally advanced rectal cancer (LARC). A total of 50 MSS LARC patients will receive 2 cycles of PD-1 antibody, followed by capecitabine plus irinotecan radiosensitized neoadjuvant chemoradiotherapy, and another 3 cycles of PD-1 antibody, finally received the total mesorectal excision (TME) and 6 cycles of adjuvant chemotherapy of XELOX. The tumor response grade, adverse effects and long-term prognosis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmed adenocarcinoma
2. clinical stage T3-4 and/or N+
3. the distance from anal verge less than 12 cm
4. without distance metastases
5. age 18-70 years old, female and male
6. KPS >=70
7. UGT1A1*28 6/6 or 6/7
8. the MSI status is MSS or p-MMR
9. without previous anti-cancer therapy or immunotherapy
10. with good compliance
11. signed the inform consent

Exclusion Criteria:

1. pregnancy or breast-feeding women
2. history of other malignancies within 5 years
3. serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
4. immunodeficiency disease or long-term using of immunosuppressive agents
5. baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
6. DPD deficiency
7. UGT1A1*28 7/7
8. the MSI status is MSI-H or d-MMR
9. allergic to any component of the therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | The pathologic complete response rate was evaluated after surgery, which was scheduled 7-8 weeks after the end of chemoradiotherapy
  Pathologic Complete Response Rate

SECONDARY OUTCOMES:
Disease free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  3 year disease free survival rate
Local recurrence free survival | From date of randomization until the date of first documented pelvic failure, assessed up to 36 months.
  3 year local recurrence free survival rate
Overall survival | From date of randomization until the date of death from any cause, assessed up to 36 months.
  3 year overall survival rate
Adverse effects | From date of randomization until the date of death from any cause, assessed up to 5 years
  Chemoradiation-related or immunotherapy-related adverse events
Surgical complications | The surgery was scheduled 7-8 weeks after the end of chemoradiotherapy. And the surgical complications were assessed up to 5 years from the surgery.
  Surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.
Performance Status (Zubrod-ECOG-WHO method), range 0-5. The higher scores mean a worse quality of life. | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated
Karnofsky Performance Status, range 0-100. The higher scores mean a better quality of life. | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated
Quality of Life Scale, range 0-60. It evaluates the quality of life from 12 aspects, including appetite, mental status, sleep quality, fatigue, etc. The higher scores mean a better quality of life. | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: zhen zhang, M.D, PH.D, Principal Investigator — Fudan University
Locations (1):
- Zhen Zhang, Shanghai, Shanghai Municipality, China